CLINICAL TRIAL: NCT02669758
Title: A Phase 3, Multicenter Study to Assess the Long Term Safety and Tolerability of ALKS 3831 in Subjects With Schizophrenia
Brief Title: A Long-Term Safety and Tolerability Study of ALKS 3831 in Adults With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK3831-A306
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
Keywords: Alkermes; ALKS 3831; Samidorphan; Schizophrenia; Safety
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 3831 (Experimental): Olanzapine + samidorphan; administered as a coated bilayer tablet.
  Interventions: Drug: ALKS 3831

INTERVENTIONS:
Drug: ALKS 3831 — Tablets were administered for daily dosing

SUMMARY:
The primary objective of this study is to evaluate the long term safety and tolerability of ALKS 3831 in subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the 4-week treatment period (all visits up to and including end of treatment visit) in the antecedent study ALK3831-A305 within 7 days.
* Agrees to use an acceptable method of contraception for the duration of the study.
* Additional criteria may apply.

Exclusion Criteria:

* Subject is currently taking medications that are contraindicated with olanzapine use.
* Subject has a positive test for drugs of abuse at study entry.
* Subject is pregnant, planning to become pregnant, or breastfeeding during the study.
* Additional criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (31):
- United States (14):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Lemon Grove, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Dallas, Texas
- Bulgaria (9):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Lovech
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Plovdiv
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Tserova Koria
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Serbia (3):
  - Alkermes Investigational Site, Belgrade
  - Alkermes Investigational Site, Kragujevac
  - Alkermes Investigational Site, Novi Kneževac
- Ukraine (5):
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Kiev
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Stepanovka
  - Alkermes Investigational Site, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who completed the 4-week treatment period of the antecedent study, ALK3831-A305, were eligible to be enrolled in Study ALK3831-A306 within 7 days of their last study visit in ALK3831-A305.
Pre-assignment Details: A total of 4 subjects enrolled but were not dosed. Three subjects were lost-to-follow-up prior to receiving study drug, and one subject was not compliant with study drug. A total of 277 patients were administered at least one dose of ALKS 3831 and were included in the safety population.
Groups:
- ALKS 3831: Administered as a coated bilayer tablet.
  ALKS 3831: Daily dosing
Period: Overall Study
Arm/Group | ALKS 3831
Started | 277
Completed | 183
Not Completed | 94
Not completed — Withdrawal by Subject | 43
Not completed — Lost to Follow-up | 19
Not completed — Adverse Event | 16
Not completed — Non-Compliance with Study Drug | 8
Not completed — Lack of Efficacy | 5
Not completed — Pregnancy | 1
Not completed — Study noncompliance | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population includes all subjects who received at least one dose of study drug.
Arm/Group | ALKS 3831
Number analyzed (Participants) | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 269
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 52
  White | 218
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: Count of participants]
  United States | 75
  Ukraine | 69
  Bulgaria | 100
  Serbia | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Up to 52 weeks
Population: Safety population includes all subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831
Number analyzed (Participants) | 277
Participants | 136

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | ALKS 3831
All-Cause Mortality (participants affected / at risk) | 0/277
Serious Adverse Events (participants affected / at risk) | 8/277
Other Adverse Events (participants affected / at risk) | 102/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 3831 (N=277)
Schizophrenia (Psychiatric disorders) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 3831 (N=277)
Weight increased (Investigations) | 37 (40)
Blood insulin increased (Investigations) | 6 (6)
Blood prolactin increased (Investigations) | 6 (6)
Weight decreased (Investigations) | 6 (6)
Somnolence (Nervous system disorders) | 23 (27)
Headache (Nervous system disorders) | 11 (13)
Anxiety (Psychiatric disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 6 (6)
Schizophrenia (Psychiatric disorders) | 6 (6)
Nasopharyngitis (Infections and infestations) | 11 (11)
Extra dose administered (Injury, poisoning and procedural complications) | 9 (11) — Resulted from the errors made by the subjects or caregivers while taking the study medication
Dry mouth (Gastrointestinal disorders) | 7 (9)
Social stay hospitalisation (Social circumstances) | 7 (7) — Per protocol social stay hospitalizations were not considered Serious Adverse Events, and were recorded as AEs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT02669758/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT02669758/SAP_001.pdf